CLINICAL TRIAL: NCT06828055
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled, 13-week Dose Finding Study of VK2735 Oral Formulation for Weight Management in Subjects Who Are Obese, or Overweight With at Least One Weight-related Comorbid Condition
Brief Title: VK2735 for Weight Management Phase 2 (Venture Oral Dosing)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Viking Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VK2735-202
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Weight Loss
Keywords: Overweight Obese
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Placebo Assignment (Placebo Comparator): VK2735 (Placebo) administered Daily
  Interventions: Drug: Placebo
- Active Assignment (Dose #1) (Experimental): VK2735 is a peptide GLP-1 and GIP dual agonist administered Daily
  Interventions: Drug: VK2735
- Active Assignment (Dose #2) (Experimental): VK2735 is a peptide GLP-1 and GIP dual agonist administered Daily
  Interventions: Drug: VK2735
- Active Assignment (Dose #3) (Experimental): VK2735 is a peptide GLP-1 and GIP dual agonist administered Daily
  Interventions: Drug: VK2735
- Active Assignment (Dose #4) (Experimental): VK2735 is a peptide GLP-1 and GIP dual agonist administered Daily
  Interventions: Drug: VK2735
- Active Assignment (Dose #5) (Experimental): VK2735 is a peptide GLP-1 and GIP dual agonist administered Daily
  Interventions: Drug: VK2735
- Active Assignment (Dose #6) (Experimental): VK2735 is a peptide GLP-1 and GIP dual agonist administered Daily
  Interventions: Drug: VK2735

INTERVENTIONS:
Drug: Placebo — Matching Placebo to VK2735
  Arms: Placebo Assignment
Drug: VK2735 — Active Treatment
  Arms: Active Assignment (Dose #1); Active Assignment (Dose #2); Active Assignment (Dose #3); Active Assignment (Dose #4); Active Assignment (Dose #5); Active Assignment (Dose #6)

SUMMARY:
This is a phase 2, 13-week randomized, double-blind, placebo-controlled, parallel arm dose-finding study that will evaluate the safety, tolerability, weight loss efficacy, pharmacodynamic effects, and pharmacokinetics of VK2735 Oral Formulation in adults who are obese (BMI ≥30 kg/m2) or who are overweight (BMI ≥27 kg/m2) with at least one weight-related co-morbid condition.

VK2735 or matched placebo will be administered once daily.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years of age at the time of signing the informed consent.
2. Body mass index (BMI) ≥30 kg/m2 OR ≥27 kg/m2 with at least one weight-related co-morbid condition (treated or untreated), and BMI <50 kg/m2

   * Weight-related co-morbid conditions include hypertension, dyslipidemia, obstructive sleep apnea or cardiovascular disease.
   * BMI calculated at the Screening visit will be used to determine eligibility.

Exclusion Criteria:

1. History of or current clinically significant medical or psychiatric disorder that, in the opinion of the Investigator, does not support study participation
2. Self-reported body weight change of 5% or more within 3 months of screening
3. Current or past diagnosis of diabetes mellitus (including type 1, type 2, gestational)
4. Current or past diagnosis of chronic pancreatitis
5. Calcitonin ≥50 ng/L measured by central laboratory at screening (individuals with elevated calcitonin at initial screening may be re-screened)
6. Any GLP-1 receptor agonist or GLP-1/GIP dual agonist within 6 months of Screening
7. Any prescription or over-the-counter medications intended for weight loss within 6 months of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2024-12-18 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Percent (relative) change from baseline in body weight after 13 weeks of treatment | 13 Weeks
  To measure the efficacy of oral VK2735 for weight loss in adult Subjects who are obese, or overweight with at least one weight-related comorbid condition

SECONDARY OUTCOMES:
Proportion of Subjects losing ≥5% and ≥10% of baseline weight at Week 13. Observed and change from baseline in body weight (kg) after 13 weeks of treatment | 13 Weeks
  To measure the efficacy of oral VK2735 for weight loss in adult Subjects who are obese, or overweight with at least one weight-related comorbid condition

OTHER OUTCOMES:
Incidence of Treatment-emergent Adverse Events, incidence of Treatment-Emergent Serious Adverse Events and incidence of Adverse Events of Special Interest | 13 Weeks
  To evaluate the safety and tolerability of oral VK2735 for weight loss in adult Subjects who are obese, or overweight with at least one weight-related comorbid condition

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Viking Clinical Site #111, Peoria, Arizona
  - Viking Clinical Site #105, Lake Forest, California
  - Viking Clinical Site #101, Clearwater, Florida
  - Viking Clinical Site #108, Largo, Florida
  - Viking Clinical Site #107, Ocoee, Florida
  - Viking Clinical Site #102, Port Orange, Florida
  - Viking Clinical Site #100, Indianapolis, Indiana
  - Viking Clinical Site #110, Louisville, Kentucky
  - Viking Clinical Site #114, Marrero, Louisiana
  - Viking Clinical Site #109, City of Saint Peters, Missouri
  - Viking Clinical Site #112, Kansas City, Missouri
  - Viking Clinical Site #113, Butte, Montana
  - Viking Clinical Site #103, Knoxville, Tennessee
  - Viking Clinical Site #104, Austin, Texas
  - Viking Clinical Site #106, San Antonio, Texas